CLINICAL TRIAL: NCT05417841
Title: A Multicenter, Randomized, Open, Parallel-controlled Clinical Trial to Compare the Efficacy and Safety of IDegAsp BID and IDegAsp QD+2IAsp in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy of Insulin Degludec/Insulin Aspart in Patients With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLD-C-21003
Record Dates: First submitted 2022-06-08; First posted 2022-06-14 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDegAsp group (Experimental): IDegAsp twice daily
  Interventions: Drug: Insulin Degludec and Insulin Aspart Injection
- IDegAsp + IAsp group (Active Comparator): IDegAsp once daily plus IAsp twice daily
  Interventions: Drug: Insulin Degludec and Insulin Aspart Injection; Drug: Insulin Aspart Injection

INTERVENTIONS:
Drug: Insulin Degludec and Insulin Aspart Injection — To evaluate the efficacy and safety of the IDegAsp BID in T2DM
  Other Names: Ryzodeg®
Drug: Insulin Aspart Injection — To evaluate the efficacy and safety of the IDegAsp QD plus IAsp BID in T2DM
  Other Names: NovoRapid®
  Arms: IDegAsp + IAsp group

SUMMARY:
In this multicenter, randomized, open-label, parallel-controlled, non-inferiority clinical trial, the efficacy and safety of insulin degludec/insulin aspart (IDegAsp) twice daily will be compared with degludec/insulin aspart (IDegAsp) once daily plus insulin aspart (IAsp) twice daily after 16weeks of treatment in patients with type 2 diabetes mellitus. This trial will enable primary assessment of the clinically relevant endpoint of a change in HbA1c.

DETAILED DESCRIPTION:
The objective of the current study is to investigate the efficacy and safety of IDegAsp twice daily compared with IDegAsp once daily plus IAsp twice daily for 16 weeks in patients with type 2 diabetes mellitus. The primary endpoint in this study is the change from baseline in HbA1c. Patients with type 2 diabetes who meet the entry criteria are planned for inclusion in this trial. Approximately 224 patients will be enrolled in the study. Patients who qualify will be randomized to IDegAsp group or IDegAsp + IAsp group. Duration of treatment includes 3-week screening period, 16-week treatment observation period and 1-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Informed consent has been obtained before any trial-related activities;
* 2. Patients aged 18~75 years old (including 18 years old and 75 years old);
* 3. Clinical diagnosis of type 2 diabetes ≥ 6 months according to WHO diagnostic criteria before screening;
* 4. Use basal insulin once a day with or without other hypoglycemic drugs for at least 3 months before randomization;
* 5. Glycated hemoglobin between 7.0%~10.0% within 3 month before randomization (including the critical value);
* 6. Body mass index (BMI)≤40.0kg/m2;

Exclusion Criteria:

* 1. Suffering from type 1 diabetes, or special type of diabetes;
* 2. Known premixed insulin or IDegAsp used 3 month before randomization;
* 3. Changes in concomitant medications that are expected to significantly interfere with glucose metabolism;
* 4. Known or suspected subjects are allergic to test drugs, excipients or related similar products and excipients;
* 5. Cardiovascular and cerebrovascular disease, defined as: congestive heart failure (NYHA class III-IV), diagnosis of unstable angina pectoris, stroke and/or myocardial infarction within 6 months before screening; or planned/coronary artery , carotid artery, peripheral artery revascularization;
* 6. According to the judgment of the investigator, repeated hypoglycemia perception impairment and severe hypoglycemia events occurred before screening;
* 7. Abnormal and clinically significant hemoglobin laboratory test results;
* 8. Hepatic insufficiency, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 times the upper limit of the normal range at screening; renal insufficiency, defined as (but not limited to) serum creatinine Levels ≥1.5mg/dL (132umol/L, men) and ≥1.4mg/dL (123umol/L, women), or massive proteinuria (>2 g/day);
* 9. Uncontrolled/untreated hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg) before randomization;
* 10. Two or more events of ketoacidosis or hyperglycemia and hyperosmolar state requiring hospitalization within 6 months prior to screening, or significant diabetic complications, such as symptomatic autonomic neuropathy, diabetic gastric mildew paralysis, proliferative retinopathy, etc. occured;
* 11. According to the judgment of the investigator, significant changes in lifestyle are expected during the trial period, such as shift work (including persistent night/evening shift work) and highly irregular diet and living habits;
* 12. Pregnant or breastfeeding women; those who have a pregnancy plan during the entire trial period and are unwilling to take one or more non-drug contraceptive measures (such as complete abstinence, contraceptive ring, partner ligation, etc.) during the trial;
* 13. Participate in any clinical trial within the past 3 months;
* 14. Those who are not suitable to participate in the trial according to the investigator's judgment, or any clinically significant disease or condition that the investigator believes may affect the results of the trial, such as: a history of hemolytic anemia or sickle cell anemia, a previous history of tumor or cancer Patients with a medical history, patients with a known history of alcohol, drug or drug abuse, blood transfusions or severe blood loss within the first 3 months of screening, or patients with poor adherence in the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
HbA1c | 16 weeks
  the change from baseline in HbA1c after 16 weeks of treatment in all patients

SECONDARY OUTCOMES:
HbA1c response | 16 weeks
  the percentage of patients with HbA1c < 7.0% in patients without definite hypoglycemia after 16 weeks of treatment
Body weight | 16 weeks
  the body weight change from baseline after 16 weeks of treatment
Fasted Blood Glucose | 16 weeks
  the change from baseline in fasting blood glucose after 16 weeks of treatment
7-Point Self-monitoring Blood Glucose | 16 weeks
  the change from baseline in 7-point self-monitoring blood glucose profile after 16 weeks of treatment
Continuous Glucose Monitoring | 14-16 weeks
  the change from Baseline in Mean Glucose of CGM at Weeks 14-16 of Treatment
Percentage of Time In Range | 14-16 weeks
  the change from Baseline in Percentage of Readings in Target Range for Blood Glucose Values at Weeks 14-16 of Treatment
Percentage of Time Below Range | 14-16 weeks
  the change from Baseline in Percentage of Readings below Target Range for Blood Glucose Values at Weeks 14-16 of Treatment
Percentage of Time Above Range | 14-16 weeks
  the change from Baseline in Percentage of Readings above Target Range for Blood Glucose Values at Weeks 14-16 of Treatment
Glucose Management Indicator | 14-16 weeks
  the change from Baseline in estimated HbA1c at Weeks 14-16 of Treatment
Glucose Variability | 14-16 weeks
  Change from Baseline in Glucose Variability (Coefficient of Variation) of CGM at Weeks 14-16 of Treatment
Time In Range | 14-16 weeks
  the change from Baseline of time in Target Range for Blood Glucose Values at Weeks 14-16 of Treatment
Time Below Range | 14-16 weeks
  the change from Baseline of time below Target Range for Blood Glucose Values at Weeks 14-16 of Treatment
Time Above Range | 14-16 weeks
  the change from Baseline of time above Target Range for Blood Glucose Values at Weeks 14-16 of Treatment

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Jilin University Sino-Japanese Friendship Hospital, Changchun, Jilin
  - The Second Affiliated Medical College of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Aerospace general hospital, Beijing
  - Beijing Boai Hospital, Beijing
  - Beijing Hospital, Beijing
  - Peking university shougang hospital, Beijing

IPD SHARING:
Plan to Share IPD: No
We plan not to make individual participant data (IPD) available to other researchers.